CLINICAL TRIAL: NCT05622318
Title: A Phase II Trial of De-escalated PTCy and Ruxolitinib for GVHD Prophylaxis in Patients Undergoing Reduced Intensity Conditioning Allogeneic HCT
Brief Title: De-escalated Cyclophosphamide (PTCy) and Ruxolitinib for Graft-versus-Host Disease (GVHD) Prophylaxis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment complete but will expand with pending amendment
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sameem M. Abedin, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00046962
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Graft-versus-host Disease
Keywords: Graft-versus-host disease; Ruxolitinib; Graft-versus-host disease prophylaxis
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide; Tacrolimus; Mycophenolic Acid; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Graft-versus-host disease prophylaxis (Experimental): Following reduced intensity conditioning and 8/8-matched peripheral blood transplant on Day 0, all patients will receive a GVHD prophylaxis post-transplant composed of the following: (i) cyclophosphamide administered at 25 mg/kg on Day +3 and +4, (ii) tacrolimus beginning on Day +5 and through Day +180 and administered with a trough target of 5-10 ng/ml through Day +90 and tapered thereafter; (iii) mycophenolate mofetil (MMF) administered at 15 mg/kg thrice daily beginning on Day +5 through Day +35; and (iv) ruxolitinib administered at 5 mg twice daily starting after engraftment (between Days +30 and +60) and continuing through one year post transplant.
  Interventions: Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Cyclophosphamide — 25 mg/kg by IV on Days +3 and +4.
  Other Names: Cytoxan
Drug: Tacrolimus — Target level 5-10 ng/mL (If the subject experiences nausea and vomiting that prevents the oral intake of tacrolimus anytime during treatment, tacrolimus is to be given by IV at the appropriate dose that was used to obtain the therapeutic level [IV:PO ratio = 1:4]). Administered Days +5 through +90. Taper after Day +90 and discontinue on Day +180.
  Other Names: Astagraf XL; Envarsus XR; Prograf
Drug: Mycophenolate Mofetil — 15 mg/kg tablet thrice daily Days +5 through +35 every eight hours.
  Other Names: CellCept
Drug: Ruxolitinib — 5 mg tablet twice daily after engraftment through Day +365. Taper after Day +365.
  Other Names: INC424; Jakafi

SUMMARY:
This is an open-label phase 2 study designed to explore the efficacy and safety of low-dose PTCy-ruxolitinib GVHD prophylaxis in older adults undergoing allogeneic HCT with a matched sibling or unrelated donor with a peripheral blood stem cell graft.

DETAILED DESCRIPTION:
Following reduced intensity conditioning and 8/8-matched peripheral blood transplant on Day 0, all patients will receive a GVHD prophylaxis post-transplant composed of the following: (i) cyclophosphamide administered at 25 mg/kg on Day +3 and +4, (ii) tacrolimus beginning on Day +5 and through Day +180 and administered with a trough target of 5-10 ng/ml through Day +90 and tapered thereafter; (iii) mycophenolate mofetil (MMF) administered at 15 mg/kg thrice daily beginning on Day +5 through Day +35; and (iv) ruxolitinib administered at 5 mg twice daily starting after engraftment (between Days +30 and +60) and continuing through one year post transplant.

ELIGIBILITY:
Inclusion Criteria:

1. History of hematologic malignancy.
2. Must be in remission:

   * Acute Leukemia, chronic leukemia, or myelodysplasia/myeloproliferative neoplasm (excluding primary myelofibrosis): No circulating blasts and <5% blasts in the bone marrow.
   * Hodgkin and non-Hodgkin lymphomas: Chemo-sensitive disease at time of transplant
3. Patients must have a related or unrelated peripheral blood stem cell donor that is an 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing. Unrelated donors must be willing to donate peripheral blood stem cells and meet NMDP criteria for donation.
4. Planned reduced intensity conditioning therapy with fludarabine/melphalan, with total dose of melphalan of 100-140 mg/m^2 IV or fludarabine/busulfan with total dose of busulfan of 6.4 mg/kg IV.
5. Karnofsky Performance Scale of 60 or greater.
6. Male participants must agree to abstinence or to use of barrier contraception during the entire study period.
7. Female participants of childbearing potential will require a negative pregnancy test and should agree to practice two effective methods of contraception during the entire study period.
8. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Prior allogeneic HCT or Chimeric antigen receptor (CAR) -T cell therapy.
2. Patients with liver dysfunction evidenced by bilirubin ≥2x upper limit normal (ULN), except for a history of Gilbert syndrome.
3. Patients with renal impairment defined by creatinine<2mg/dL.
4. Patients with cardiac dysfunction defined by a left ventricular ejection fraction ≤45%.
5. Patients with pulmonary dysfunction defined by a forced expiratory volume in the first second (FEV1) or diffusing capacity for carbon monoxide (DLCO) (corrected for hemoglobin) ≤50% of predicted.
6. Patients with a chronic or active infection requiring systemic treatment during and after transplant.
7. Presence of other active malignant disease diagnosed within 12 months, except for adequately treated non-melanoma skin cancer, adequately treated melanoma grade 2 or less, or cervical intraepithelial neoplasia. Active malignancy is malignancy receiving treatment.
8. Pregnant or lactating subjects.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
The number of subjects who experience GVHD-free survival. | One year (365 Days) after hematopoietic cell transplantation (HCT)
  This measure is defined as being alive without having experienced grade III/IV acute GVHD, or chronic GVHD requiring systemic immune suppression.

SECONDARY OUTCOMES:
The number of subjects with acute GVHD at Day +100. | Day +100 after HCT
  The staging and grading of acute GVHD will be done according to Consensus GVHD grading criteria.
The number of subjects with acute GVHD at Day +180. | Day +180 after HCT
  The staging and grading of acute GVHD will be done according to Consensus GVHD grading criteria.
The number of subjects with chronic GVHD at one year. | One year after HCT
  Chronic GVHD will be graded as mild, moderate, or severe according to the NIH consensus criteria.
The number of subjects with non-relapse mortality at Day +100. | Day +100 after HCT
  This is defined as death before day +100 after transplant that was not preceded by recurrent or progressive malignancy.
The number of subjects with non-relapse mortality at one year. | One year after HCT
  This is defined as death before day +100 after transplant that was not preceded by recurrent or progressive malignancy.
Overall survival at one year. | One year after HCT
  This is defined as the number of subjects alive one year after HCT.

CONTACTS AND LOCATIONS:
Overall Officials: Sameem Abedin, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No